CLINICAL TRIAL: NCT02212080
Title: One-center, Randomized, Placebo-controlled, Double Blind, Parallel Group Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single Oral Doses (5-1000 mg, Solution) of BAY1214784 Including the Relative Bioavailability of BAY1214784 Administered as Solution With Two Different Concentrations in 56 Healthy Postmenopausal Women
Brief Title: First in Human Study in Healthy Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of BAY1214784
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16924; 2014-000412-34 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Clinical Trials, Phase I as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY1214784 (Experimental): Dose 1 to 7 of BAY1214784
  Interventions: Drug: BAY1214784
- Placebo (Placebo Comparator): Placebo Dose 1 to 7 of BAY1214784
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1214784 — Escalating doses of 5, 20, 60, 150, 300, 600, 1000 mg of BAY1214784; single dose administration; liquid dosage form
  Arms: BAY1214784
Drug: Placebo — Dose 1, 2,3, 4, 5, 6 and 7 of respective placebos; single dose administration; liquid dosage form
  Arms: Placebo

SUMMARY:
This study is a first in human study that will investigate the safety, tolerability and pharmacokinetics of ascending single doses of BAY1214784 using a placebo controlled, randomized, single center design. In addition the bioavailability of two different liquid formulations will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Age 45 to 65 years
* Body mass index (BMI) above/equal 20 and below/equal 30 kg/m2
* Postmenopausal state

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known or suspected malignant or benign tumors
* Known or suspected liver disorders, relevant kidney diseases, known cardiovascular diseases, known metabolic disorders
* Regular use of medicines

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Up to 2 weeks after dosing
Severity of adverse events (mild, moderate, severe) | Up to 2 weeks after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Mönchengladbach, North Rhine-Westphalia
  - Erfurt, Thuringia